CLINICAL TRIAL: NCT04218942
Title: Interest of Rocamed Urethral Device for Treatment of Acute or Chronic Urinary Retention in Males
Brief Title: Rocamed Urethral Device (RUD) and Urinary Retention in Males
Acronym: RUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0395
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Urinary Retention
Keywords: Urethral Device; Foley catheterization
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective non randomised feasibility study (Experimental)
  Interventions: Device: Exime is the name of the single use temporary prostatic stent used instead of the Foley catheter

INTERVENTIONS:
Device: Exime is the name of the single use temporary prostatic stent used instead of the Foley catheter — Insertion after instillation of a local lubricant anesthetic gel in the urethra like for Foley insertion. Calibration of the urethral meatus with a 22F Bougie. Insertion of the Bougie until abutment against the posterior wall of the bulbous urethra just below the striated sphincter. Note depth of abutment on the scale of the Bougie. Retrieve the Bougie and glide the device to the same depth until abutment against the posterior wall of the bulbous urethra. At this stage the stent is correctly positioned. Stent release: unlock the Luer connection between pusher tube and stylet . Retrieve pusher tube, stylet and flattener tube.
  Control of correct positioning: ask patient to stand up to verify the absence of any urine leak. Ask patient to void immediately to control clear urine output.

SUMMARY:
Prospective non randomized study of the feasibility of the insertion of Rocamed urethral device by hand manipulation, i.e., without use of cystoscopy, sonography or fluoroscopy. Patients with an acute urinary retention treated by Foley catheterization in the Emergency department have a few days later a trial of Foley removal in the ambulatory unit of the Urology department. In case of failure of the Foley removal trial, i.e., recurrence of urinary retention, patients will be proposed either the insertion of a new Foley or insertion of the urethral device. After signature of an informed consent, insertion of the urethral device will be performed after instillation in the urethra of a local anesthetic gel. Device insertion success rate and complications will be studied. The device will be left in place for one month. Tolerance and complications during the month with the device in place will be studied. At one month the device will be removed: the ease of retrieval of the device and complications will be studied. Patient and doctor satisfaction with the urethral device will be compared to patient and doctor satisfaction with the Foley.

ELIGIBILITY:
Inclusion Criteria:

* Male > 18 years old
* Acute retention treated by Foley
* Failure of Foley removal trial
* Clear urine
* No urinary infection
* Efficient striated sphincter

Exclusion Criteria:

* Urethral stenosis
* Hematuria macroscopic
* Urinary infection
* Anticoagulant treatment
* Lidocaine allergy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in whom the device will be inserted only by hand manipulation | Day 0

SECONDARY OUTCOMES:
Patient tolerance during device insertion: analogic visual scale 0-10 (0 : no pain / 10 : worst pain imaginable) | Day 0 (Day of device insertion)
Patient tolerance during one month: analogic visual scale 0-10 (0 : excellent tolerance / 10 : intolerable) | 1 Month
Flowmetry with device in place ml/sec | Day 0 (Day of device insertion)
Patient tolerance during retrieval of the device : analogic visual scale 0-10 (0 : no pain / 10 : worst pain imaginable) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Urologie Hôpital Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite, France